CLINICAL TRIAL: NCT01191697
Title: Phase II Trial of CAPOX, Bevacizumab and Trastuzumab for Patients With HER2-Positive Metastatic Esophagogastric Cancer
Brief Title: CAPOX, Bevacizumab and Trastuzumab for Patients With HER2-Positive Metastatic Esophagogastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Peter Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-457
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Results first posted 2023-09-05 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: HER2 positive
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Bevacizumab; Trastuzumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine (Experimental): Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine for patients with HER2-positive metastatic esophagogastric cancer. Each cycle is 21 days.
  Cycle 1, Day 1 Trastuzumab (loading dose) 4mg/kg IV
  Cycle 2, Day 1 and all Subsequent Cycles Bevacizumab (7.5mg/kg) IV Trastuzumab (6mg/kg) IV Oxaliplatin (130mg/m2) IV Capecitabine (1200mg/m2) PO (taken Days 1-14 of each cycle)
  Patients remained on treatment until disease progression, intercurrent illness that prevented further administration of treatment, unacceptable adverse events, participant decision to withdraw consent or general or specific changes in the participant's condition that rendered the participant unacceptable for further treatment.
  Interventions: Drug: bevacizumab; Drug: trastuzumab; Drug: oxaliplatin; Drug: capecitabine

INTERVENTIONS:
Drug: bevacizumab — Given intravenously on day 1 of each cycle beginning cycle 2
  Other Names: Avastin
Drug: trastuzumab — Given intravenously on day 1 of each treatment cycle
  Other Names: Herceptin
Drug: oxaliplatin — Given intravenously on day one of each cycle beginning cycle 2
Drug: capecitabine — Taken orally on days 1-14 of each cycle beginning cycle 2
  Other Names: xeloda

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a combination of chemotherapy, capecitabine and oxaliplatin, plus the antibodies bevacizumab and trastuzumab. Trastuzumab (also called Herceptin) is an antibody that attacks HER2 protein in tumor cells. Bevacizumab (also called Avastin) works by slowing or stopping the growth of cells in cancer tumors by decreasing the blood supply of the tumors. If blood supply is decreased, oxygen and nutrients that are needed for tumor growth are decreased. The chemotherapy used in this trial is called CAPOX, which is an abbreviation of capecitabine and oxaliplatin.

DETAILED DESCRIPTION:
* We recommend that the participants have a vascular access device, more commonly known as a PORT, inserted prior to starting chemotherapy. A port is a small device that is inserted under the skin (usually near the collar bone) by a minor surgical procedure and is then connected to one of the large veins inside the chest. The port will be used to give the intravenous medications.
* During the first cycle, the participant will receive trastuzumab intravenously on Day 1. Cycle 2 will then start one week later. On this day, bevacizumab will be given intravenously first followed by trastuzumab and then oxaliplatin. The participant will then start taking capecitabine tablets orally twice a day for 14 days. Each treatment cycle is 21 days long.
* Participants will have the following tests and procedures at specific time points during study treatment; physical exam, blood tests, CT scan, MUGA scan or echocardiogram, and urine test.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HER2-positive esophageal, GE junction or gastric adenocarcinoma that is metastatic or unresectable.
* All patients must have available tumor sample (either paraffin block or 15 freshly cut, unstained slides) prior to study entry.

Part II: Patient must have primary esophagogastric tumor in place or other tumor that is accessible for mandatory biopsy.

* Measurable disease, defined in RECIST 1.1
* 18 years of age or older
* Life expectancy of greater than 12 weeks
* ECOG performance status of 0 or 1
* Organ and marrow function as outlined in the protocol
* Women of child-bearing potential and men must agree to use adequate contraception during study participation and for 30 days from the date of the last study drug administration.
* Part II only: Participant agrees to undergo mandatory pre and post loading dose of trastuzumab biopsy for correlative science.

Exclusion Criteria:

* Prior therapy with any of the following; capecitabine, oxaliplatin, bevacizumab or trastuzumab is not allowed. May have received and completed adjuvant therapy at least 6 months prior to study entry or one prior therapy for metastatic disease as long as it did not include any of the above agents.
* Chemotherapy or radiotherapy to greater then 25% of bone marrow within 4 weeks prior to entering the study.
* Palliative radiation therapy to isolated bone metastasis within 2 weeks of initiating therapy.
* Major surgery, open biopsy, significant traumatic injury within 4 weeks prior to study entry,.
* Minor surgery, including placement of vascular access device within 7 days prior to the first dose of bevacizumab.
* Residual toxicity from prior chemotherapy and/or radiation therapy of Grade 2 or greater.
* Participants may not be receiving any concurrent investigational agents
* Active brain or other CNS metastasis by history or clinical examination.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine, bevacizumab or trastuzumab. No known allergy or hypersensitivity to Chinese hamster ovary, or any of the study agents. No known DPD deficiency.
* Warfarin is prohibited; anticoagulation using low molecular weight heparin is allowed.
* Uncontrolled, intercurrent illness
* Patients with a history of other malignancy are not eligible except for the following circumstances: disease-free for at least 3 years and are deemed to be at low risk for recurrence of that malignancy; cervical cancer in situ, basal cell or squamous cell carcinoma of the skin that was treated with curative intent within the past 5 years.
* Known HIV seropositivity, hepatitis C, acute or chronic hepatitis B or other serious active infection
* LVEF less than 50% as determined by MUGA scan or echocardiogram within 28 days prior to initiation of therapy
* Inadequately controlled hypertension
* History of prior hypertensive crisis or hypertensive encephalopathy
* History of any arterial thrombosis, CVA, TIA, MI or unstable angina in past 6 months.
* Evidence of bleeding diathesis or coagulopathy
* Serious, unhealed wounds, bone fractures or skin ulcers
* Pregnant or breast feeding
* Greater than grade 1 peripheral neuropathy at baseline
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2024-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Pohl H, Welch HG. The role of overdiagnosis and reclassification in the marked increase of esophageal adenocarcinoma incidence. J Natl Cancer Inst. 2005 Jan 19;97(2):142-6. doi: 10.1093/jnci/dji024. PMID 15657344
- [Background] Cancer Genome Atlas Research Network; Analysis Working Group: Asan University; BC Cancer Agency; Brigham and Women's Hospital; Broad Institute; Brown University; Case Western Reserve University; Dana-Farber Cancer Institute; Duke University; Greater Poland Cancer Centre; Harvard Medical School; Institute for Systems Biology; KU Leuven; Mayo Clinic; Memorial Sloan Kettering Cancer Center; National Cancer Institute; Nationwide Children's Hospital; Stanford University; University of Alabama; University of Michigan; University of North Carolina; University of Pittsburgh; University of Rochester; University of Southern California; University of Texas MD Anderson Cancer Center; University of Washington; Van Andel Research Institute; Vanderbilt University; Washington University; Genome Sequencing Center: Broad Institute; Washington University in St. Louis; Genome Characterization Centers: BC Cancer Agency; Broad Institute; Harvard Medical School; Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University; University of North Carolina; University of Southern California Epigenome Center; University of Texas MD Anderson Cancer Center; Van Andel Research Institute; Genome Data Analysis Centers: Broad Institute; Brown University:; Harvard Medical School; Institute for Systems Biology; Memorial Sloan Kettering Cancer Center; University of California Santa Cruz; University of Texas MD Anderson Cancer Center; Biospecimen Core Resource: International Genomics Consortium; Research Institute at Nationwide Children's Hospital; Tissue Source Sites: Analytic Biologic Services; Asan Medical Center; Asterand Bioscience; Barretos Cancer Hospital; BioreclamationIVT; Botkin Municipal Clinic; Chonnam National University Medical School; Christiana Care Health System; Cureline; Duke University; Emory University; Erasmus University; Indiana University School of Medicine; Institute of Oncology of Moldova; International Genomics Consortium; Invidumed; Israelitisches Krankenhaus Hamburg; Keimyung University School of Medicine; Memorial Sloan Kettering Cancer Center; National Cancer Center Goyang; Ontario Tumour Bank; Peter MacCallum Cancer Centre; Pusan National University Medical School; Ribeirao Preto Medical School; St. Joseph's Hospital &Medical Center; St. Petersburg Academic University; Tayside Tissue Bank; University of Dundee; University of Kansas Medical Center; University of Michigan; University of North Carolina at Chapel Hill; University of Pittsburgh School of Medicine; University of Texas MD Anderson Cancer Center; Disease Working Group: Duke University; Memorial Sloan Kettering Cancer Center; National Cancer Institute; University of Texas MD Anderson Cancer Center; Yonsei University College of Medicine; Data Coordination Center: CSRA Inc.; Project Team: National Institutes of Health. Integrated genomic characterization of oesophageal carcinoma. Nature. 2017 Jan 12;541(7636):169-175. doi: 10.1038/nature20805. Epub 2017 Jan 4. PMID 28052061
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Background] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- [Background] Andrulis IL, Bull SB, Blackstein ME, Sutherland D, Mak C, Sidlofsky S, Pritzker KP, Hartwick RW, Hanna W, Lickley L, Wilkinson R, Qizilbash A, Ambus U, Lipa M, Weizel H, Katz A, Baida M, Mariz S, Stoik G, Dacamara P, Strongitharm D, Geddie W, McCready D. neu/erbB-2 amplification identifies a poor-prognosis group of women with node-negative breast cancer. Toronto Breast Cancer Study Group. J Clin Oncol. 1998 Apr;16(4):1340-9. doi: 10.1200/JCO.1998.16.4.1340. PMID 9552035
- [Background] Bartley AN, Washington MK, Colasacco C, Ventura CB, Ismaila N, Benson AB 3rd, Carrato A, Gulley ML, Jain D, Kakar S, Mackay HJ, Streutker C, Tang L, Troxell M, Ajani JA. HER2 Testing and Clinical Decision Making in Gastroesophageal Adenocarcinoma: Guideline From the College of American Pathologists, American Society for Clinical Pathology, and the American Society of Clinical Oncology. J Clin Oncol. 2017 Feb;35(4):446-464. doi: 10.1200/JCO.2016.69.4836. Epub 2016 Nov 14. PMID 28129524
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Tabernero J, Hoff PM, Shen L, Ohtsu A, Shah MA, Cheng K, Song C, Wu H, Eng-Wong J, Kim K, Kang YK. Pertuzumab plus trastuzumab and chemotherapy for HER2-positive metastatic gastric or gastro-oesophageal junction cancer (JACOB): final analysis of a double-blind, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2018 Oct;19(10):1372-1384. doi: 10.1016/S1470-2045(18)30481-9. Epub 2018 Sep 11. PMID 30217672
- [Background] Zhao D, Klempner SJ, Chao J. Progress and challenges in HER2-positive gastroesophageal adenocarcinoma. J Hematol Oncol. 2019 May 17;12(1):50. doi: 10.1186/s13045-019-0737-2. PMID 31101074
- [Background] Janjigian YY, Kawazoe A, Yanez P, Li N, Lonardi S, Kolesnik O, Barajas O, Bai Y, Shen L, Tang Y, Wyrwicz LS, Xu J, Shitara K, Qin S, Van Cutsem E, Tabernero J, Li L, Shah S, Bhagia P, Chung HC. The KEYNOTE-811 trial of dual PD-1 and HER2 blockade in HER2-positive gastric cancer. Nature. 2021 Dec;600(7890):727-730. doi: 10.1038/s41586-021-04161-3. Epub 2021 Dec 15. PMID 34912120
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Ohtsu A, Shah MA, Van Cutsem E, Rha SY, Sawaki A, Park SR, Lim HY, Yamada Y, Wu J, Langer B, Starnawski M, Kang YK. Bevacizumab in combination with chemotherapy as first-line therapy in advanced gastric cancer: a randomized, double-blind, placebo-controlled phase III study. J Clin Oncol. 2011 Oct 20;29(30):3968-76. doi: 10.1200/JCO.2011.36.2236. Epub 2011 Aug 15. PMID 21844504
- [Background] Cleary JM, Horick NK, McCleary NJ, Abrams TA, Yurgelun MB, Azzoli CG, Rubinson DA, Brooks GA, Chan JA, Blaszkowsky LS, Clark JW, Goyal L, Meyerhardt JA, Ng K, Schrag D, Savarese DMF, Graham C, Fitzpatrick B, Gibb KA, Boucher Y, Duda DG, Jain RK, Fuchs CS, Enzinger PC. FOLFOX plus ziv-aflibercept or placebo in first-line metastatic esophagogastric adenocarcinoma: A double-blind, randomized, multicenter phase 2 trial. Cancer. 2019 Jul 1;125(13):2213-2221. doi: 10.1002/cncr.32029. Epub 2019 Mar 26. PMID 30913304
- [Background] Fuchs CS, Shitara K, Di Bartolomeo M, Lonardi S, Al-Batran SE, Van Cutsem E, Ilson DH, Alsina M, Chau I, Lacy J, Ducreux M, Mendez GA, Alavez AM, Takahari D, Mansoor W, Enzinger PC, Gorbounova V, Wainberg ZA, Hegewisch-Becker S, Ferry D, Lin J, Carlesi R, Das M, Shah MA; RAINFALL Study Group. Ramucirumab with cisplatin and fluoropyrimidine as first-line therapy in patients with metastatic gastric or junctional adenocarcinoma (RAINFALL): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):420-435. doi: 10.1016/S1470-2045(18)30791-5. Epub 2019 Feb 1. PMID 30718072
- [Background] Van Cutsem E, de Haas S, Kang YK, Ohtsu A, Tebbutt NC, Ming Xu J, Peng Yong W, Langer B, Delmar P, Scherer SJ, Shah MA. Bevacizumab in combination with chemotherapy as first-line therapy in advanced gastric cancer: a biomarker evaluation from the AVAGAST randomized phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2119-27. doi: 10.1200/JCO.2011.39.9824. Epub 2012 May 7. PMID 22565005
- [Background] Laughner E, Taghavi P, Chiles K, Mahon PC, Semenza GL. HER2 (neu) signaling increases the rate of hypoxia-inducible factor 1alpha (HIF-1alpha) synthesis: novel mechanism for HIF-1-mediated vascular endothelial growth factor expression. Mol Cell Biol. 2001 Jun;21(12):3995-4004. doi: 10.1128/MCB.21.12.3995-4004.2001. PMID 11359907
- [Background] Konecny GE, Meng YG, Untch M, Wang HJ, Bauerfeind I, Epstein M, Stieber P, Vernes JM, Gutierrez J, Hong K, Beryt M, Hepp H, Slamon DJ, Pegram MD. Association between HER-2/neu and vascular endothelial growth factor expression predicts clinical outcome in primary breast cancer patients. Clin Cancer Res. 2004 Mar 1;10(5):1706-16. doi: 10.1158/1078-0432.ccr-0951-3. PMID 15014023
- [Background] Singh R, Kim WJ, Kim PH, Hong HJ. Combined blockade of HER2 and VEGF exerts greater growth inhibition of HER2-overexpressing gastric cancer xenografts than individual blockade. Exp Mol Med. 2013 Nov 1;45(11):e52. doi: 10.1038/emm.2013.111. PMID 24176949
- [Background] Liu K, Chen H, You Q, Shi H, Wang Z. The siRNA cocktail targeting VEGF and HER2 inhibition on the proliferation and induced apoptosis of gastric cancer cell. Mol Cell Biochem. 2014 Jan;386(1-2):117-24. doi: 10.1007/s11010-013-1850-0. Epub 2013 Oct 26. PMID 24158524
- [Background] Adalsteinsson VA, Ha G, Freeman SS, Choudhury AD, Stover DG, Parsons HA, Gydush G, Reed SC, Rotem D, Rhoades J, Loginov D, Livitz D, Rosebrock D, Leshchiner I, Kim J, Stewart C, Rosenberg M, Francis JM, Zhang CZ, Cohen O, Oh C, Ding H, Polak P, Lloyd M, Mahmud S, Helvie K, Merrill MS, Santiago RA, O'Connor EP, Jeong SH, Leeson R, Barry RM, Kramkowski JF, Zhang Z, Polacek L, Lohr JG, Schleicher M, Lipscomb E, Saltzman A, Oliver NM, Marini L, Waks AG, Harshman LC, Tolaney SM, Van Allen EM, Winer EP, Lin NU, Nakabayashi M, Taplin ME, Johannessen CM, Garraway LA, Golub TR, Boehm JS, Wagle N, Getz G, Love JC, Meyerson M. Scalable whole-exome sequencing of cell-free DNA reveals high concordance with metastatic tumors. Nat Commun. 2017 Nov 6;8(1):1324. doi: 10.1038/s41467-017-00965-y. PMID 29109393
- [Background] Pectasides E, Stachler MD, Derks S, Liu Y, Maron S, Islam M, Alpert L, Kwak H, Kindler H, Polite B, Sharma MR, Allen K, O'Day E, Lomnicki S, Maranto M, Kanteti R, Fitzpatrick C, Weber C, Setia N, Xiao SY, Hart J, Nagy RJ, Kim KM, Choi MG, Min BH, Nason KS, O'Keefe L, Watanabe M, Baba H, Lanman R, Agoston AT, Oh DJ, Dunford A, Thorner AR, Ducar MD, Wollison BM, Coleman HA, Ji Y, Posner MC, Roggin K, Turaga K, Chang P, Hogarth K, Siddiqui U, Gelrud A, Ha G, Freeman SS, Rhoades J, Reed S, Gydush G, Rotem D, Davison J, Imamura Y, Adalsteinsson V, Lee J, Bass AJ, Catenacci DV. Genomic Heterogeneity as a Barrier to Precision Medicine in Gastroesophageal Adenocarcinoma. Cancer Discov. 2018 Jan;8(1):37-48. doi: 10.1158/2159-8290.CD-17-0395. Epub 2017 Oct 4. PMID 28978556
- [Background] Grillo F, Fassan M, Sarocchi F, Fiocca R, Mastracci L. HER2 heterogeneity in gastric/gastroesophageal cancers: From benchside to practice. World J Gastroenterol. 2016 Jul 14;22(26):5879-87. doi: 10.3748/wjg.v22.i26.5879. PMID 27468182
- [Background] Zhang L, Hamdani O, Gjoerup O, Cho-Phan C, Snider J, Castellanos E, Nimeiri H, Frampton G, Venstrom JM, Oxnard G, Klempner SJ, Schrock AB. ERBB2 Copy Number as a Quantitative Biomarker for Real-World Outcomes to Anti-Human Epidermal Growth Factor Receptor 2 Therapy in Advanced Gastroesophageal Adenocarcinoma. JCO Precis Oncol. 2022 Jan;6:e2100330. doi: 10.1200/PO.21.00330. PMID 35050711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 61 participants assessed for eligibility, 37 met the inclusion criteria and enrolled for treatment. One patient withdrew consent prior to starting therapy. 36 were evaluable for efficacy and safety.
Period: Overall Study
Arm/Group | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine
Started | 37
Analyzed Popopulation | 36 (1 participant withdrew consent prior to starting threapy.)
Completed | 0
Not Completed | 37
Not completed — Death | 1
Not completed — Physician Decision | 2
Not completed — Pursue chemoradiation | 2
Not completed — Break from chemotherapy | 2
Not completed — Withdrawal by Subject | 1
Not completed — Surveillance | 1
Not completed — Adverse Event | 2
Not completed — Subject never received treatment and wasn't analyzed. | 1
Not completed — Not completed but analyzed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 55.5 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Patients received a median of 19 cycles of therapy (Interquartile range (IQR): 8 - 34.5 cycles). Median duration of follow-up of 23.2 months (IQR: 11.0 - 46.9 months ).
Measure: Number; unit: percentage of patients
Arm/Group | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine
Number analyzed (Participants) | 36
percentage of patients | 81

2. Secondary Outcome: Median Overall Survival
Description: Overall survival based on the Kaplan-Meier method is defined as the time from randomization to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Time Frame: 23.2 months (IQR: 11.0 - 46.9 months ).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine
Number analyzed (Participants) | 36
months | 23.2 [16.6 to 36.4]

3. Secondary Outcome: Median Duration of Response (DOR)
Description: DOR is defined as the time from date of first documented confirmed objective response to date of first documented progressive disease (PD). Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: 23.2 months (IQR: 11.0 - 46.9 months ).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine
Number analyzed (Participants) | 29
months | 14.9 [2.4 to 95.9]

4. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Patients received a median of 19 cycles of therapy (Interquartile range (IQR): 8 - 34.5 cycles). Median duration of follow up of 23.2 months (IQR: 11.0 - 46.9 months ).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine
Number analyzed (Participants) | 36
months | 14.0 [11.3 to 36.4]

ADVERSE EVENTS:
Time Frame: All adverse events experienced by participants will be collected from the time of the first dose of study treatment, throughout the study, and until the final study visit. Participants continuing to experience toxicity at the off-study visit may be contacted for additional assessments until the toxicity has resolved or is deemed irreversible. (10 years and 7 months)
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Per the source vocabulary (CTCAEv4.0) there is a category "Other, specify" for each system organ class. No further data is available to specify classification beyond this general term.
Arm/Group | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine
All-Cause Mortality (participants affected / at risk) | 31/36
Serious Adverse Events (participants affected / at risk) | 13/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine (N=36)
Dehydration (Metabolism and nutrition disorders) | 5
Pulmonary Embolism (Blood and lymphatic system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hponatremia (Blood and lymphatic system disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Hypertriglyceridemia (Blood and lymphatic system disorders) | 1
Perforated Gallbladder (Gastrointestinal disorders) | 1
Hernia (General disorders) | 1
Cardiac Arrest/Arrhythmia (Cardiac disorders) | 1
GE Junction Bleed (Gastrointestinal disorders) | 1
Mental Status Changed (Psychiatric disorders) | 1
Leptomeningeal Carcinomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fatal Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal Bleed (Gastrointestinal disorders) | 1
Fracture (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab, Bevacizumab, Oxaliplatin and Capecitabine (N=36)
Anemia (Blood and lymphatic system disorders) | 26
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3
heart failure (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 29
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (gastric pneumatosis) (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 27
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 4
Rectal hemorrhage (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 13
Fatigue (General disorders and administration site conditions) | 13
Pain (General disorders and administration site conditions) | 4
Chills (General disorders and administration site conditions) | 1
Fatigue (General disorders and administration site conditions) | 16
Fever (General disorders and administration site conditions) | 3
Gait disturbance (General disorders and administration site conditions) | 1
Infusion related reaction (General disorders and administration site conditions) | 6
Neck edema (General disorders and administration site conditions) | 1
Non-cardiac chest pain (General disorders and administration site conditions) | 1
Pain (General disorders and administration site conditions) | 3
Hepatobiliary disorders - Other (hepatic abscess) (Hepatobiliary disorders) | 1
Gallbladder infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Paronychia (Infections and infestations) | 5
Rhinitis infective (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 14
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 19
Blood bilirubin increased (Investigations) | 6
CD4 lymphocytes decreased (Investigations) | 1
Creatinine increased (Investigations) | 3
Ejection fraction decreased (Investigations) | 2
Investigations - Other (altered mental status) (Investigations) | 1
Investigations - Other, specify (Investigations) | 8
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 21
Weight loss (Investigations) | 8
White blood cell decreased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 3
Dysesthesia (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 7
Memory impairment (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 32
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Proteinuria (Renal and urinary disorders) | 11
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 10
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 2
Nail loss (Skin and subcutaneous tissue disorders) | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 15
Thromboembolic event (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT01191697/Prot_SAP_000.pdf